CLINICAL TRIAL: NCT05358873
Title: A Phase I Double-blind, Randomized, Placebo-controlled Study to Evaluate Safety of Hypromellose-based Nasal Spray Solution Containing Human IgG1 Anti-SARS-CoV-2 Antibody Cocktail in Healthy Volunteers
Brief Title: Efficacy and Safety of Nasal Spray Solution Containing Human IgG1 Anti-COVID-19 Antibody Cocktail
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Collaborators: Ramathibodi Hospital (Other); Ever Medical Technology Co., Ltd. (Unknown); The Government Pharmaceutical Organization (Other Government); Ministry of Health, Thailand (Other Government); HIBIOCY CO., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: DMS-001/2565
Record Dates: First submitted 2022-04-27; First posted 2022-05-03 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-04

CONDITIONS: SARS CoV 2 Infection; SARS-CoV-2 Acute Respiratory Disease
Keywords: SARS-CoV-2; SARS-CoV-2 inhibition; Nasal Spray; Anti-SARS-CoV-2; Antibody Cocktail
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Tolerability and safety of the study product will be evaluated when given 3 times a day for 7 days in 36 healthy volunteers.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Human IgG1 anti-SARS-CoV-2 antibody cocktail (Experimental): Subjects will receive the Hypromellose-based nasal spray solution containing human IgG1 anti-SARS-CoV-2 antibody cocktail (i.e., applied into both nostrils by spraying two times per nostril) 3 times a day from Day 1 to Day 7. Each day the study products will be self-administered at 8 am, 2 pm, and 8 pm.
  Interventions: Device: Human IgG1 anti-SARS-CoV-2 antibody cocktail
- Placebo (Placebo Comparator): Subjects will receive the Normal saline solution (0.9% NaCl) nasal spray solution containing human IgG1 anti-SARS-CoV-2 antibody cocktail (i.e., applied into both nostrils by spraying two times per nostril) 3 times a day from Day 1 to Day 7. Each day the study products will be self-administered at 8 am, 2 pm, and 8 pm.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Human IgG1 anti-SARS-CoV-2 antibody cocktail — Hypromellose-based nasal spray solution containing human IgG1 anti-SARS-CoV-2 antibody cocktail
  Arms: Human IgG1 anti-SARS-CoV-2 antibody cocktail
Device: Placebo — Normal saline
  Arms: Placebo

SUMMARY:
Hypromellose-based nasal spray solution containing human IgG1 anti-SARS-CoV-2 antibody cocktail is a medical device innovated to provide the dual-action physical barrier on nasal mucosa that aids the natural defence in which the mucus layer is fortified by a steric barrier-forming agent HPMC and invading viral particles of all major SARS-CoV-2 VOCs, including Delta and Omicron, are locally trapped and blocked from entering the cells by the highly-specific human IgG1 anti-SARS-CoV-2 monoclonal antibody cocktail.

DETAILED DESCRIPTION:
The transmission of SARS-CoV-2 through inhalation results in the nasal cavity and nasopharynx being the primary entry point of the virus and containing the highest viral load in the body during the virus incubation period. Recently, the administration of vaccines and agents via a nasal route has gained a lot of momentum because it takes advantage of the direct delivery of an agent to the site of primary infection. The local defence system, especially antibody-mediated immunity at the nasal epithelium, is crucial for COVID-19 prevention. However, people who responded to the vaccination against COVID-19 typically maintain sufficient local antibody levels in the nasal cavity for only a short period; hence a repeated boosting strategy is required to control the rate of SARS-CoV-2 breakthrough infection. In addition, the new VOCs such as Omicron are known to escape vaccine immunity; therefore, an innovative approach is needed in this unprecedented situation

Hypromellose-based nasal spray solution containing human IgG1 anti-SARS-CoV-2 antibody cocktail is a medical device innovated to provide the dual-action physical barrier on nasal mucosa that aids the natural defence in which the mucus layer is fortified by a steric barrier-forming agent HPMC and invading viral particles of all major SARS-CoV-2 VOCs, including Delta and Omicron, are locally trapped and blocked from entering the cells by the highly-specific human IgG1 anti-SARS-CoV-2 monoclonal antibody cocktail.

ELIGIBILITY:
Inclusion criteria

1. Male or female, ≥ 18 and ≤ 50 years of age with BMI ≥ 18 and ≤ 30 kg/m2
2. Healthy as defined by:

   1. No previous clinically significant disease and surgery within 4 weeks prior to dosing.
   2. No previous sinus and nasal septum surgery or radiotherapy
   3. No evidence of clinically significant history of neurological, endocrine, cardiovascular, pulmonary, hematological, immunologic, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease which the Investigator believes may be detrimental to the study or its aims.
   4. No evidence of febrile or infectious disease within 1 week prior to dosing.
3. Have received at least 2 doses of COVID-19 vaccine.
4. Have no history of close contact with COVID-19 patients within 2 weeks before enrolment
5. Have negative result of COVID-19 test using RT-PCR method using sample collected from nasopharyngeal or nasal or oropharyngeal swab within 72 hours before sinusoscopy
6. Provide signed written informed consent prior to the initiation of any study-specific procedures.
7. Willing and able to comply with the requirements of the protocol and be available for the planned duration of the trial.

Exclusion criteria

1. Any clinically significant abnormality at physical examination at screening or enrolment
2. Vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 40 or over 90 mmHg, heart rate less than 40 or over 100 bpm, respiratory rate less than 10 or over 22 bpm, oral temperature less than 35.5°C or over 37.5°C) at screening.
3. Positive urine pregnancy test for women or women who are breast feeding
4. History of COVID-19 infection within 3 months before enrollment
5. History of allergic reactions or hypersensitivity to any excipients of the study products.
6. Use any nasal product use within 14 days prior to the first dosing
7. History of pulmonary infiltrate or pneumonia within 6 months before the screening visit.
8. Signs or symptoms of respiratory tract abnormalities such as allergies or chronic obstructive pulmonary disease.
9. History or signs of chronic allergic rhinitis that may interfere with study procedures and/or interpretation of local adverse events.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Adverse events | 1 Day
  Tolerability and safety of the study product as measured by treatment emergent adverse events (TEAEs)

SECONDARY OUTCOMES:
Percentage of inhibition against SAR-CoV-2 in the nasal fluid | 14 Days
  SARS-CoV-2 inhibition property of the study product as measured by the percentage of inhibition against SAR-CoV-2 in the nasal fluid before and after the study product application via cPass™ SARS-CoV-2 Neutralization Antibody Detection Kit

OTHER OUTCOMES:
Sino-Nasal Outcome Test-22 (SNOT-22) | 14 Days
  Subject will be asked to respond to the SNOT-22 every day during enrolment to the end-of-study visit. The SNOT-22 is a validated 22-item CRS-specific QoL instrument which is scored where 0="No problem", 1="Very mild problem", 2="Mild or slight problem", 3="Moderate problem", 4="Severe problem", and 5="Problem as bad as it can be
Total Nasal Symptom Score (TNSS) Questionnaire | 14 Days
  Subject will be asked to respond to the TNSS questionnaire every day during enrolment to the end-of-study visit. Total nasal symptoms score (TNSS) is a brief questionnaire which evaluate the severity of main symptoms of allergic rhinitis. It consists of three questions which assess nasal obstruction, itching/sneezing and secretion/runny nose.

CONTACTS AND LOCATIONS:
Overall Officials: Thanarathi Imsuwansr, MD, Principal Investigator — National Cancer Institute, Thailand; Dhammika Leshan Wannigama, MD PhD, Study Director — Chulalongkorn University; Thitinan Jongthitinon, MD, Study Chair — National Cancer Institute, Thailand
Locations (1):
- National Cancer Institute of Thailand, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Imsuwansri T, Jongthitinon T, Pojdoung N, Meesiripan N, Sakarin S, Boonkrai C, Wongtangprasert T, Phakham T, Audomsun T, Attakitbancha C, Saelao P, Muanwien P, Tian MT, Tongchusak S, Sangruji B, Wannigama DL, Sawangmake C, Rodprasert W, Le QD, Purbantoro SD, Vasuntrarak K, Nantavisai S, Sirilak S, Uppapong B, Sapsutthipas S, Trisiriwanich S, Somporn T, Usoo A, Mingngamsup N, Phumiamorn S, Aumklad P, Arunprasert K, Patrojanasophon P, Opanasopit P, Pesirikan N, Nitisaporn L, Pitchayakorn J, Narkthong T, Mahong B, Chaiyo K, Srisutthisamphan K, Viriyakitkosol R, Aeumjaturapat S, Jongkaewwattana A, Bunnag S, Pisitkun T. Assessment of safety and intranasal neutralizing antibodies of HPMC-based human anti-SARS-CoV-2 IgG1 nasal spray in healthy volunteers. Sci Rep. 2023 Sep 20;13(1):15648. doi: 10.1038/s41598-023-42539-7. PMID 37730833